CLINICAL TRIAL: NCT00787631
Title: Analysis of Immunological Reactions to Pollen-Related Foods in Birch Pollen-Allergic Patients
Brief Title: Analysis of Immunological Reactions to Foods in Birch Pollen-Allergic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Tamar Kinaciyan, MD, Ass. Prof., DIAID, Dep. of Dermatology, MUV
Other Study IDs: TK01/2008
Record Dates: First submitted 2008-10-23; First posted 2008-11-07 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-10

CONDITIONS: Allergic Rhinitis; Food Allergy
Keywords: birch pollen pollen allergy; oral allergy syndrome to apple; cross reactivity; bet v 1; mal d 1
MeSH Terms: conditions — Rhinitis, Allergic; Food Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A high number of birch pollen-allergic individuals develop hypersensitivity reactions to certain foods, e.g. apples. This food allergy is due to immunological cross-reactivity. Birch pollen-related foods contain proteins, e.g. Mal d 1 in apple, that are structurally related with the major birch pollen allergen, Bet v 1. Hence IgE antibodies and T lymphocytes specific for Bet v 1 recognize these food proteins which results in activation of the immune system and, consequently, in clinical symptoms.

In the present study the investigators intend to investigate if and how the consumption of birch pollen-related food allergens affects birch pollen allergy. In other words, the investigators are interested to analyse whether Bet v 1-related food allergens activate Bet v 1-specific memory cells and thus, contribute to the maintenance of the pollen allergy outside the pollen season. Data obtained in this study will help to clarify the immunological and clinical role of cross-reactivity between pollen and food allergies and will reveal whether avoidance of such foods should be recommended for the patients. Finally, novel approaches for diagnosis and therapy of pollen-related food allergens can be developed.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy birch pollen allergic (rhinoconjunctivitis)persons
* Positive SPT and RAST to birch pollen
* Sensitized to Bet v 1

Exclusion Criteria:

* Persons suffering from malignancies, autoimmune and cardiopulmonary diseases
* Anemia
* Hyper-IgE syndrome
* Treatment with ß-blockers, permanent treatment with antihistaminics, leucotriene antagonists, corticosteroids

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: otherwise healthy birch pollen allergic (rhinoconjunctivitis)persons suffering also from oral allergy syndrome to apple.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-01 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Kinaciyan, Ass Prof MD, Principal Investigator — Dept. of Dermatology, Medical University of Vienna